CLINICAL TRIAL: NCT01363661
Title: Double-blind Parallel Placebo-controlled Study to Evaluate the Effect of Molsidomine on the Endothelial Dysfunction in Patients With Stable Angina Pectoris Undergoing a Percutaneous Coronary Intervention
Brief Title: Effect of Molsidomine on the Endothelial (Internal Layer of Blood Vessels) Dysfunction in Patients With Angina Pectoris
Acronym: MEDCOR
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Therabel Pharma SA/NV (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MEDCOR 2011; 2011-000190-31 (EudraCT Number)
Record Dates: First submitted 2011-04-01; First posted 2011-06-01 (Estimated); Results first posted 2014-09-26 (Estimated); Last update posted 2014-10-06 (Estimated); Status verified 2014-09

CONDITIONS: Stable Angina Pectoris; Atherosclerosis
Keywords: angina pectoris; atherosclerosis; endothelial dysfunction
MeSH Terms: conditions — Angina, Stable; Atherosclerosis; Angina Pectoris | interventions — Molsidomine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Molsidomine (Experimental): Coruno (molsidomine 16 mg tablet; per os; once daily)
  Interventions: Drug: Coruno
- Placebo (Placebo Comparator): Placebo (16 mg tablet; once a day)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Coruno — Molsidomine 16 mg tablet, per os, once a day
  Other Names: Molsidomine
  Arms: Molsidomine
Drug: Placebo — Placebo (16 mg tablet, per os; once-daily)
  Arms: Placebo

SUMMARY:
Molsidomine used as an add-on treatment on standard care therapy should be superior to placebo used also as an add-on treatment on standard care therapy on improving the endothelial function (endothelium score measured by reactive hyperemia - peripheral arterial tonometry [RH-PAT]) after 12 months of treatment in patients with stable angina patients and undergoing elective percutaneous coronary intervention.

The study will be double-blind, parallel-group, randomised, multicentre, sequential, placebo-controlled study.

The device used to determine RH-PAT will be EndoPAT. Duration of the treatment = one year.

DETAILED DESCRIPTION:
A Data Steering Committee (DSC) will blindly assess the recruitment rate, the variability of RH-PAT within and between centres, and the safety on a regular basis.

Sequential approach:

* In the first phase (Phase A) of the study, 180 patients will be enrolled in order to get at least 50 completers after 12 months of treatment. A statistical evaluation of the primary endpoint will be done by an Independent Biostatistician after approximately 50 patients have completed the study in accordance with the protocol.
* The results will be examined by an Independent Data Monitoring Committee (IDMC)which will assess the results and advise the sponsor as to:

  1. Continue the study if the primary objective has not been achieved but the difference between the two groups is at least 10% (difference considered clinically significant). In this case, the sample size will be recalculated by the Independent Biostatistician taking into account actual difference and variability. The total number of patients to be enrolled in addition in Phase B will be calculated with precision. Depending on IDMC recommendations, the number of investigating centres will be increased or not for Phase B. If the right number of patients has already been enrolled, Phase B will not start. The study will stop when all enrolled patients have completed the one-year treatment period.
  2. Terminate the study, if the difference between the two groups is less than 10%.
  3. Consider the study as completed if the primary endpoint has been achieved.

Treatment allocation: Balanced allocation between molsidomine and placebo (1:1) with a stratification for consumption of statins, for the type of stent (drug-eluting stent or bare-metal) and for consumption of angiotensin-converting enzyme inhibitors (ACEIs).

Data collection: Electronic Case Report Form (eCRF).

Duration of study: A minimum of 30 months (16 months for inclusion and 14 months for the study) for Phase A.

Number of investigational centres:

* Up to 10 centres for Phase A
* To be determined for Phase B based on Phase A.

ELIGIBILITY:
Inclusion Criteria:

* Aged at least 18 years.
* No treatment with molsidomine and/or long-acting nitrates (oral or patches) for more than 48 hours during the month preceding percutaneous coronary intervention (PCI) and no treatment with these same drugs within 3 days before PCI.
* Patients who the investigator believes that they and/or their Legally Acceptable Representative (LAR) can and will comply with the requirements of the protocol.
* Written informed consent from the patient or from the LAR.
* Patients who underwent PCI for stable angina pectoris one month prior to the start of the study.
* Patients presenting endothelial dysfunction at Month 0 (score of the Endo-PAT <0.40).

Exclusion Criteria:

* Pre-menopausal women.
* Patient with a clinically-active malignancy.
* Known major renal insufficiency or known significant hepatic insufficiency.
* History of psychological disorder, mental dysfunction, alcohol or drug abuse or any other factor which might interfere with the ability to cooperate in the study.
* Participation in another clinical trial which has not yet reached its primary endpoint or with the same primary endpoint during the previous month.
* Concurrently participating in another clinical study, at any time during the study period, in which the subject will be exposed to an investigational or a non-investigational product (vaccine, drug or device).
* Hypersensitivity to molsidomine or to one of its excipients.
* Peri-procedural infarction: creatine kinase-muscle/brain (CK-MB) >3 times the upper reference limit.
* Clinically significant abnormal pre-PCI CK-MB and troponin: any elevation above the upper reference limit.
* Intolerance to galactose, deficiency in Lapp lactase or glucose-galactose malabsorption.
* Left ventricular insufficiency (New York Heart Association [NYHA] class III or IV) with an ejection fraction <35%.
* Acute circulatory insufficiency (e.g. cardiogenic shock).
* Hypotension: systolic blood pressure <100 mmHg and/or diastolic blood pressure <70 mmHg.
* Atrial fibrillation
* Acute myocardial infarction during the preceding month.
* Unsuccessful PCI: residual stenosis of at least 50%.
* Patient taking phosphodiesterase-5 inhibitors, such as sildenafil (Viagra®), vardenafil (Levitra®) and tadalafil (Cialis®)
* Patient taking nebivolol (Nobiten®)
* Patient taking ibuprofen + L-arginine as excipient (Spidifen®)
* Patient meeting any contraindication(s) from Coruno®. Please refer to Coruno® (molsidomine 16 mg o.d.)Summary of Product Characteristics (SPC).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 165 (Actual)
Dates: Start 2011-06; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Emanuele Barbato, MD, Principal Investigator — Cardiology Center, Onze Lieve Vrouw Ziekenhuis Aalst
Locations (1):
- Onze Lieve Vrouw Ziekenhuis, Aalst, Belgium

REFERENCES:
- [Background] Barbato E, Herman A, Benit E, Janssens L, Lalmand J, Hoffer E, Chenu P, Guedes A, Missault L, Pirenne B, Cardinal F, Vercauteren S, Wijns W. Double-blind parallel placebo-controlled study to evaluate the effect of molsidomine on the endothelial dysfunction in patients with stable angina pectoris undergoing percutaneous coronary intervention: the MEDCOR Trial. J Cardiovasc Transl Res. 2014 Mar;7(2):226-31. doi: 10.1007/s12265-013-9513-9. Epub 2013 Oct 19. PMID 24142804
- [Derived] Barbato E, Herman A, Benit E, Janssens L, Lalmand J, Hoffer E, Chenu P, Guedes A, Missault L, Pirenne B, Cardinal F, Vercauteren S, Wijns W. Long-term effect of molsidomine, a direct nitric oxide donor, as an add-on treatment, on endothelial dysfunction in patients with stable angina pectoris undergoing percutaneous coronary intervention: results of the MEDCOR trial. Atherosclerosis. 2015 Jun;240(2):351-4. doi: 10.1016/j.atherosclerosis.2015.03.045. Epub 2015 Apr 7. PMID 25875387

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The drop-out rate post-PCI was high (>60%) mainly because the Endoscore was frequently above the pre-defined threshold post-PCI, attesting of the absence of endothelial dysfunction. Post-randomization drop-out rate was also high, 25% of patients being lost between randomization and month 12, mainly for non-serious adverse events.
Period: Overall Study
Arm/Group | Molsidomine | Placebo
Started | 32 | 32
Completed | 18 | 28
Not Completed | 14 | 4
Not completed — Adverse Event | 9 | 2
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Protocol Violation | 1 | 0
Not completed — Lost to Follow-up | 3 | 1

BASELINE CHARACTERISTICS:
Population: This population corresponded to the per protocol cohort: patients who had been randomized to placebo or molsidomine and who had completed the study in accordance with the protocol.
Groups:
- Total: Total of all reporting groups
Arm/Group | Molsidomine | Placebo | Total
Number analyzed (Participants) | 18 | 28 | 46
Age, Continuous [Mean (Standard Deviation); unit: Years] | 62.4 (10.2) | 64.1 (9.9) | 63.5 (9.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 5 | 7
  Male | 16 | 23 | 39
Region of Enrollment [Number; unit: participants]
  Belgium | 18 | 28 | 46

OUTCOME MEASURES:

1. Primary Outcome: Change Versus Baseline in the Score of the EndoPAT in the Two Groups After One Year of Treatment (Month 12).
Description: The results are expressed mean relative change (%) between month 12 and baseline. A positive result means improvement in the score of the EndoPAT between baseline and month 12. It could be considered as a surrogate of a decrease of the endothelial dysfunction. A negative percentage means the inverse. The are no fixed limits to the scale. The minimum observed was -275% and the maximum observed was +4200%.
Time Frame: 12 months
Population: Per protocol population
Measure: Mean (Standard Deviation); unit: Relative change versus baseline (%)
Arm/Group | Molsidomine | Placebo
Number analyzed (Participants) | 18 | 28
Relative change versus baseline (%) | 330.60 (1014.98) | 164.08 (433.41)

2. Secondary Outcome: Change Versus Baseline in the Score of the EndoPAT in the Two Groups After Six Months of Treatment (Month 6).
Description: The results are expressed mean relative change (%) between month 6 and baseline. A positive result means improvement in the score of the EndoPAT between baseline and month 6. It could be considered as a surrogate of a decrease of the endothelial dysfunction. A negative percentage means the inverse. The are no fixed limits to the scale. The minimum observed was -200% and the maximum observed was +6100%.
Time Frame: Month 6
Population: Per protocol population
Measure: Mean (Standard Deviation); unit: Relative change versus baseline (%)
Arm/Group | Molsidomine | Placebo
Number analyzed (Participants) | 18 | 28
Relative change versus baseline (%) | 361.98 (1248.52) | 326.26 (1155.90)

3. Secondary Outcome: Change Versus Baseline in the Augmentation Index in the Two Groups After Six and Twelve Months of Treatment (Months 6 and 12).
Description: The results are expressed mean relative change (%) between month 6 or month 12, and baseline. A positive result means improvement in the augmentation index between baseline and month 6 or month 12. It could be considered as a surrogate of a decrease of the arterial stiffness. A negative percentage means the inverse. The are no fixed limits to the scale. At month 6,the minimum observed was -139% and the maximum observed was +1600%.At month 12, the minimum observed was -524% and the maximum observed was +1600%.
Time Frame: Month 6 and Month 12
Population: Per protocol population
Measure: Mean (Standard Deviation); unit: Relative change versus baseline (%)
Arm/Group | Molsidomine | Placebo
Number analyzed (Participants) | 18 | 28
Relative change versus baseline (%)
  Month 6 | 218.07 (437.38) | 96.35 (323.14)
  Month 12 | 98.57 (470.39) | 95.13 (290.41)

4. Secondary Outcome: Change Versus Baseline in Some Specific Endothelial Biomarkers After Twelve Months of Treatment (Month 12).
Time Frame: Month 12
Population: Per protocol population
Measure: Mean (Standard Deviation); unit: Relative change versus baseline (%)
Arm/Group | Molsidomine | Placebo
Number analyzed (Participants) | 18 | 28
Relative change versus baseline (%)
  Endothelial microparticles | -40 (75) | -40 (42)
  Platelet microparticles | 0.5 (101) | -23 (252)
  Leukocyte microparticles | -39 (83) | -37 (29)
  sICAM-1 | -6 (51) | 6 (47)
  IL-8 | 13 (43) | -25 (149)
  hs-CRP | -50 (237) | -35 (163)
  MOX-LDL | 11 (80) | 41 (83)
  MPO antigen | -1 (19) | -32 (128)
  MPO activity | -43 (51) | 8 (149)
  MPO activity/antigen ratio | -42 (60) | 7 (68)

5. Secondary Outcome: Frequency of Serious Cardiovascular Events (SCEs) in the Two Groups After Twelve Months of Treatment (Month 12).
Description: Sum of the events collected during 12 months.
Time Frame: Month 12
Population: Intention-to-treat population
Measure: Number; unit: Number of events
Arm/Group | Molsidomine | Placebo
Number analyzed (Participants) | 32 | 32
Number of events | 3 | 1

6. Secondary Outcome: Frequency of AEs and SAEs in the Two Groups After Twelve Months of Treatment (Month 12).
Description: Sum of the events collected during 12 months.
Time Frame: Month 12
Population: Intention-to-treat population
Measure: Number; unit: Number of events
Arm/Group | Molsidomine | Placebo
Number analyzed (Participants) | 32 | 32
Number of events
  Non-serious AE | 57 | 79
  SAE | 7 | 12

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Molsidomine | Placebo
Serious Adverse Events (participants affected / at risk) | 7/32 | 11/32
Other Adverse Events (participants affected / at risk) | 16/32 | 22/32
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Molsidomine (N=32) | Placebo (N=32)
Acute coronary syndrome (Cardiac disorders) | 1 (1) | 0 (0)
Angina pectoris (Cardiac disorders) | 1 (1) | 1 (1)
Angina unstable (Cardiac disorders) | 2 (2) | 0 (0)
Arteriogram coronary (Cardiac disorders) | 1 (1) | 1 (1)
Bowen's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Colitis ulcerative (Gastrointestinal disorders) | 0 (0) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Epididymitis (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Haemorrhoids (Gastrointestinal disorders) | 1 (1) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Melanoma recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Myocardial ischaemia (Cardiac disorders) | 0 (0) | 1 (1)
Oesophagitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Road traffic accident (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Scapula fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Sleep study (Investigations) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Molsidomine (N=32) | Placebo (N=32)
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 4 (4)
Chest pain (Cardiac disorders) | 2 (2) | 10 (10)
Dizziness (Nervous system disorders) | 3 (3) | 1 (1)
Headache (Nervous system disorders) | 8 (8) | 3 (3)
Nasopharyngitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 4 (4)

LIMITATIONS AND CAVEATS:
Too limited sample size. Huge variability in all measurements. High drop-out rate. Add-on treatment was a challenge to demonstrate a difference between Coruno and placebo.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less